CLINICAL TRIAL: NCT04516772
Title: Post-Approval Study of the Visian Toric Implantable Collamer Lens
Brief Title: STAAR Visian Toric ICL Post-Approval Study
Acronym: TICL-PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Staar Surgical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP18-02
Record Dates: First submitted 2020-08-10; First posted 2020-08-18 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Myopic Astigmatism
Keywords: nearsightedness; phakic IOL; Toric ICL; TICL; TMICL; Visian; astigmatism
MeSH Terms: conditions — Astigmatism; Myopia

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will undergo phakic eye surgery to have the STAAR Visian Toric Implantable Collamer Lens (TICL) implanted in one or both eligible eyes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Visian TICL (Other): STAAR Visian Toric implantable collamer lens (TICL) for the correction or reduction of myopia with astigmatism.
  Interventions: Device: Visian TICL

INTERVENTIONS:
Device: Visian TICL — The Visian TICL is intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior capsule of the human crystalline lens.
  Other Names: Visian Toric ICL; TMICL

SUMMARY:
The objective of this study is to evaluate the long term (i.e. 24 months) clinical performance of the Visian® Toric Implantable Collamer® Lens (ICL).

DETAILED DESCRIPTION:
This study will be conducted at 6-8 clinical sites in the US, by surgeons qualified by experience and training to implant Visian Toric ICLs.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to high myopia with astigmatism correctable with available TICL powers.
* Stable refractive history within 0.50 D each cylinder and spherical equivalent (SE) for 1 year prior to implantation.
* Able and willing to return for scheduled follow-up examinations after surgery.
* Able to read, understand and provide written informed consent on the Institutional Review Board (IRB)-approved informed consent form (ICF) and provide authorization as appropriate for local privacy regulations.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Insulin-dependent diabetes or diabetic retinopathy.
* History of previous ocular surgery.
* Cataract of any grade.
* Monocular.
* Pregnant or nursing women, or those who plan to become pregnant over the course of this clinical study.
* Other protocol-specified exclusion criteria may apply.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Change in axis orientation of the TICL | 18 to 24 months postoperative
  Rotation of the TICL of less than or equal to five degrees in 90% of treated eyes between 18 and 24 months postoperative

SECONDARY OUTCOMES:
Absolute Rotation of the TICL in treated eyes | 1 day, 1 week, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months after surgery
  * Absolute rotation of the TICL between visits
  * Absolute rotation of the TICL <5 degrees, <10 degrees, <20 degrees, and <30 degrees from intended orientation
  * Absolute rotation of the TICL at each visit
Manifest refraction spherical equivalence (MRSE) and cylinder | 1 week, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months after surgery
  MRSE and cylinder in treated eyes
Ocular (adverse events) AEs | Through study completion, an average of 24 months
  Incidence of AEs in treated eyes

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Egamino, PhD, Study Director — VP, Clinical Affairs
Locations (8):
- United States (8):
  - Aloha Laser Vision, LLC, Honolulu, Hawaii
  - Price Vision Group,, Indianapolis, Indiana
  - Solomon Eye Physicians and Surgeons/Bowie Vision Institute, Bowie, Maryland
  - Vance Thompson Vision, Omaha, Nebraska
  - Vance Thompson Vision, West Fargo, North Dakota
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Key-Whitman Eye Center, Dallas, Texas
  - Hoopes Vision/Hoopes, Durrie, Rivera Research, Draper, Utah

IPD SHARING:
Plan to Share IPD: No